CLINICAL TRIAL: NCT04452669
Title: Double-blind, Placebo Controlled Study to Assess the Efficacy and Safety of VentaProst (Inhaled Epoprostenol Delivered Via Dedicated Delivery System) in Subjects With COVID-19 Requiring Mechanical Ventilation
Brief Title: VentaProst in Subjects With COVID-19 Requiring Mechanical Ventilation
Acronym: VPCOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerogen Pharma Limited (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APC-VPCOV-CLN-001
Record Dates: First submitted 2020-06-29; First posted 2020-06-30 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: COVID-19; ARDS
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled study comparing study treatment group to placebo controls who received SOC
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Treatment (Experimental): Up to 10 days of inhaled epoprostenol delivered by a breath actuated dedicated delivery system for patients with COVID-19 who are mechanically ventilated.
  Interventions: Drug: VentaProst (inhaled epoprostenol delivered via a dedicated delivery system)
- Placebo Control (Placebo Comparator): Up to 10 days of inhaled 0.9% sodium chloride solution delivered by a breath actuated dedicated delivery system for patients with COVID-19 who are mechanically ventilated.
  Interventions: Drug: VentaProst (inhaled epoprostenol delivered via a dedicated delivery system)

INTERVENTIONS:
Drug: VentaProst (inhaled epoprostenol delivered via a dedicated delivery system) — VentaProst delivered for up to 10 days via mechanical ventilation at a dose range that may be up or down titrated to a patient's clinical condition.
  Other Names: inhaled Flolan

SUMMARY:
The purpose of this study is to investigate whether inhaled epoprostenol given via a breath actuated delivery system will help improve oxygen levels and treatment outcomes in patients with COVID-19 who are on mechanical ventilation.

DETAILED DESCRIPTION:
This study will evaluate the potential therapeutic benefit of VentaProst in treating patients with COVID-19 at risk for respiratory and/ or cardiac/circulatory failure. This is a double-blind, placebo controlled study of VentaProst in 10 confirmed COVID-19 patients compared to 10- COVID-19 placebo patients to assess the efficacy and safety of VentaProst given over 10 days at varying doses.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 positive by RT-PCR test
* Patients who require invasive mechanical ventilation.
* Consent or professional consent obtained

Exclusion Criteria:

* Patients on ECMO support.
* Patients receiving another inhalation research medication or inhaled nitric oxide.
* Not expected to survive for 48 hours.
* Allergy to Epoprostenol and its diluent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Franco, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Treatment | Placebo Control
Started | 6 | 5
Completed | 5 | 1
Not Completed | 1 | 4
Not completed — Death | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Treatment | Placebo Control | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 3 | 2 | 5
  >65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Respiratory Failure
Description: Number of participants that were extubated
Time Frame: 10 days post-randomization
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Study Treatment | Placebo Control
Number analyzed (Participants) | 6 | 5
Participants | 3 | 2

2. Primary Outcome: Change in Cardiac/Circulatory Failure
Description: Number of participants that required ECMO or left ventricular assist device (LVAD)
Time Frame: 10 days post-randomization
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Study Treatment | Placebo Control
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from randomization through 28 days post-randomization.
Arm/Group | Study Treatment | Placebo Control
All-Cause Mortality (participants affected / at risk) | 1/6 | 4/5
Serious Adverse Events (participants affected / at risk) | 1/6 | 4/5
Other Adverse Events (participants affected / at risk) | 0/6 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment (N=6) | Placebo Control (N=5)
Worsening of ARDS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Worsening of Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hypercapnic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment (N=6) | Placebo Control (N=5)
Hypotension (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT04452669/Prot_SAP_000.pdf